CLINICAL TRIAL: NCT02985541
Title: Multi-center, Open-label, Uncontrolled Study to Assess Contraceptive Efficacy and Safety of Mirena During Extended Use Beyond 5 Years in Women 18 to 35 Years of Age Including a Subgroup Evaluation of Treatment Effect on Heavy Menstrual Bleeding
Brief Title: Mirena Extension Trial
Acronym: MET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18649
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Contraception
Keywords: Birth Control; Heavy menstrual bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Levonorgestrel IUS (Mirena, BAY86-5028) (Experimental): Mirena during extended use (Years 6 to 8).
  Interventions: Drug: Levonorgestrel IUS (Mirena, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel IUS (Mirena, BAY86-5028) — Levonorgestrel (LNG) intrauterine delivery system (IUS) with an initial in vitro release rate of 20 μg levonorgestrel per day.

SUMMARY:
The study is performed to assess if Mirena is effective and safe as a birth control method beyond 5 years of use. Further the menstrual blood loss (in women that had Mirena inserted for the indication heavy menstrual bleeding [HMB]) and safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Women, 18 to 35 years of age at the time of screening (visit 1) who are currently using Mirena for contraception or for contraception and heavy menstrual bleeding. The duration of use of the current Mirena has to be at least 4 years 6 months at the start of screening phase but not more than 5 years at visit 2 and the woman is willing to continue with its use and has a continuing need for contraception.
* Normal or clinically insignificant cervical smear not requiring further follow up

Exclusion Criteria:

* Menopausal symptoms with Follicle-stimulating hormone>30 mIU/ml
* Pregnancy or suspicion of pregnancy
* Uterine bleeding of unknown etiology
* Untreated acute cervicitis or vaginitis or other lower genital tract infections
* Increased susceptibility to pelvic infection
* Acute pelvic inflammatory disease (PID) or a history of PID unless successfully treated and which, in the investigator's opinion, has not negatively affected subject's fertility
* Congenital or acquired uterine anomaly if it distorts the uterine cavity
* History of, diagnosed or suspected genital or other malignancy and untreated cervical dysplasia
* Any active acute liver disease or liver tumor (benign or malignant)
* Clinically significant endometrial polyp(s)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 364 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (47):
- United States (47):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Encinitas, California
  - San Francisco, California
  - Ventura, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Idaho Falls, Idaho
  - Fort Wayne, Indiana
  - Newburgh, Indiana
  - Frederick, Maryland
  - Pikesville, Maryland
  - Boston, Massachusetts
  - Saginaw, Michigan
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Lawrenceville, New Jersey
  - Neptune City, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Port Jefferson, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Franklin, Ohio
  - Mayfield Heights, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Chattanooga, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Draper, Utah
  - Midlothian, Virginia
  - North Chesterfield, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 364 women entered treatment period. Of these, 2 women were not valid for FAS (full analysis set)/SAF (safety analysis set)/PAS(primary analysis set) due to incomplete source data verification.
Period: Overall Study
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Started | 364
Valid for FAS | 362
Continued Into Year 7 of Mirena Use | 305
Continued Into Year 8 of Mirena Use | 243
Completed | 223
Not Completed | 141
Not completed — Withdrawal by Subject | 33
Not completed — Lost to Follow-up | 26
Not completed — Adverse Event | 27
Not completed — Physician Decision | 2
Not completed — Pregnancy | 2
Not completed — Wish for pregnancy | 44
Not completed — Other reason | 5
Not completed — Not valid for analysis | 2

BASELINE CHARACTERISTICS:
Population: FAS (full analysis set)
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Number analyzed (Participants) | 362
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41
  Not Hispanic or Latino | 319
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 51
  White | 273
  More than one race | 14
  Unknown or Not Reported | 13
Parity [Number; unit: Participants]
  Nulliparous | 171
  Parous | 191

OUTCOME MEASURES:

1. Primary Outcome: Number of Pregnancies Per 100 Women Years (Pearl Index [PI]) Within Years 6 Thru 8 of Mirena Use
Description: The Pearl Index (PI) is defined as the number of pregnancies per 100 women years. The 3-year PI (Years 6 to 8) was obtained by dividing the number of pregnancies the occurred during that time (starting at Day 1 Year 6 and up to Day 365 of Year 8) by the time (in 100 women years) that the women were at risk of getting pregnant during that time.
Time Frame: Years 6 to 8 of Mirena use
Population: All women in the full analysis set (FAS) with an age of 33 years or younger at baseline visit (i.e. an age of 36 or younger at end of year 8).
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 women years
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Number analyzed (Participants) | 346
Pregnancies per 100 women years | 0.28 [0.03 to 1.00]
Statistical Analysis 1: Comparison: Levonorgestrel IUS (Mirena, BAY86-5028); Cumulative failure rate (Kaplan-Meier) during Years 6-8; Test type: Other; 3-year probability of getting pregnant = 0.68, 95% CI 2-sided [0.17 to 2.71]

2. Secondary Outcome: Menstrual Blood Loss (MBL) During a 30-day Period Starting at the Baseline Visit and at the End of Years 6, 7 and 8
Description: Menstrual blood loss (MBL) during a 30-day period starting at the baseline visit and at the end of Year 6, Year 7, and Year 8, measured by the alkaline hematin method. The assessment of this variable was restricted to women who had Mirena inserted for heavy menstrual bleeding (HMB).
Time Frame: Baseline and end of Years 6, 7 and 8 of Mirena use
Population: Women who had Mirena inserted for HMB
Measure: Median (Full Range); unit: mL/30 days
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Number analyzed (Participants) | 6
mL/30 days
  Beginning of Year 6 (baseline): number analyzed (Participants) | 5
  Beginning of Year 6 (baseline) | 0.000 [0.00 to 2.32]
  End of Year 6: number analyzed (Participants) | 4
  End of Year 6 | 0.000 [0.00 to 0.00]
  End of Year 7: number analyzed (Participants) | 3
  End of Year 7 | 0.000 [0.00 to 0.00]
  End of Year 8: number analyzed (Participants) | 4
  End of Year 8 | 0.000 [0.00 to 0.00]

3. Secondary Outcome: Number of Participants With Menstrual Blood Loss (MBL) (>= 80 ml Per 30 Days) at End of Year 6, 7 and 8 of Mirena Use
Description: Categorized menstrual blood loss (MBL) (≥ 80 mL per 30 days) at end of Year 6, Year 7, and Year 8. The assessment of this variable was restricted to women who had Mirena inserted for HMB.
Time Frame: At end of Year 6, 7 and 8 of Mirena use
Population: Women who had Mirena inserted for HMB
Measure: Number; unit: Participants
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Number analyzed (Participants) | 6
Participants
  End of Year 6: number analyzed (Participants) | 4
  End of Year 6 | 0
  End of Year 7: number analyzed (Participants) | 3
  End of Year 7 | 0
  End of Year 8: number analyzed (Participants) | 4
  End of Year 8 | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence (ie any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation subject after providing written informed consent for participation in the study. Serious adverse event (SAE) was defined as any untoward medical occurrence that, at any dose 1) resulted in death, 2) was life-threatening, 3) required inpatient hospitalization or prolongation of existing hospitalization, 4) resulted in persistent or significant disability/incapacity, 5) was a congenital anomaly/birth defect, or 6) was another medically important serious event as judged by the investigator. Treatment-emergent adverse event (TEAE) was defined as an AE that occurred on Day 1 Year 6 of Mirena use or later.
Time Frame: Years 6 to 8 of Mirena use
Population: Safety analysis set (SAF): All women who completed the baseline visit of the study, analyzed for the FAS.
Measure: Number; unit: Participants
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Number analyzed (Participants) | 362
Participants
  Any AE | 249
  Any SAE | 14

5. Other Pre Specified Outcome: Total LNG Concentrations in Plasma Estimated Based on the Final 8-year Population Pharmacokinetics (popPK) Model
Description: A population pharmacokinetic (popPK) analysis was performed including sparse data from the study.
Time Frame: At the beginning of Year 6 (baseline) and at the end of Years 6, 7, and 8 of Mirena use
Population: Concentrations were estimated for women who had Mirena still in place.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/L
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Number analyzed (Participants) | 361
ng/L
  At the beginning of Year 6 (baseline) | 123 (38.3)
  At the end of Year 6: number analyzed (Participants) | 330
  At the end of Year 6 | 114 (38.7)
  At the end of Year 7: number analyzed (Participants) | 275
  At the end of Year 7 | 106 (39.2)
  At the end of Year 8: number analyzed (Participants) | 224
  At the end of Year 8 | 100 (39.9)

6. Other Pre Specified Outcome: Participant's Satisfaction With Mirena by Visit
Description: Participants were asked to evaluate their satisfaction with Mirena on a 5-point scale as very satisfied, somewhat satisfied, neither satisfied or dissatisfied, dissatisfied or very dissatisfied.
Time Frame: Baseline, at end of Year 6, 7 and 8 of Mirena use
Population: Full analysis set (FAS): All women who completed the baseline visit of the study.
Measure: Number; unit: Participants
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
Number analyzed (Participants) | 362
Participants
  Baseline (very satisfied) | 342
  Baseline (somewhat satisfied) | 20
  Baseline (neither satisfied nor dissatisfied) | 0
  Baseline (dissatisfied) | 0
  Baseline (very dissatisfied) | 0
  Year 6 (very satisfied): number analyzed (Participants) | 302
  Year 6 (very satisfied) | 279
  Year 6 (somewhat satisfied): number analyzed (Participants) | 302
  Year 6 (somewhat satisfied) | 20
  Year 6 (neither satisfied nor dissatisfied): number analyzed (Participants) | 302
  Year 6 (neither satisfied nor dissatisfied) | 3
  Year 6 (dissatisfied): number analyzed (Participants) | 302
  Year 6 (dissatisfied) | 0
  Year 6 (very dissatisfied): number analyzed (Participants) | 302
  Year 6 (very dissatisfied) | 0
  Year 7 (very satisfied): number analyzed (Participants) | 243
  Year 7 (very satisfied) | 218
  Year 7 (somewhat satisfied): number analyzed (Participants) | 243
  Year 7 (somewhat satisfied) | 20
  Year 7 (neither satisfied nor dissatisfied): number analyzed (Participants) | 243
  Year 7 (neither satisfied nor dissatisfied) | 1
  Year 7 (dissatisfied): number analyzed (Participants) | 243
  Year 7 (dissatisfied) | 3
  Year 7 (very dissatisfied): number analyzed (Participants) | 243
  Year 7 (very dissatisfied) | 1
  Year 8 (very satisfied): number analyzed (Participants) | 223
  Year 8 (very satisfied) | 207
  Year 8 (somewhat satisfied): number analyzed (Participants) | 223
  Year 8 (somewhat satisfied) | 13
  Year 8 (neither satisfied nor dissatisfied): number analyzed (Participants) | 223
  Year 8 (neither satisfied nor dissatisfied) | 3
  Year 8 (dissatisfied): number analyzed (Participants) | 223
  Year 8 (dissatisfied) | 0
  Year 8 (very dissatisfied): number analyzed (Participants) | 223
  Year 8 (very dissatisfied) | 0

ADVERSE EVENTS:
Time Frame: Years 6 to 8 of Mirena use
Arm/Group | Levonorgestrel IUS (Mirena, BAY86-5028)
All-Cause Mortality (participants affected / at risk) | 0/362
Serious Adverse Events (participants affected / at risk) | 14/362
Other Adverse Events (participants affected / at risk) | 107/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levonorgestrel IUS (Mirena, BAY86-5028) (N=362)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Uterine perforation (Injury, poisoning and procedural complications) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 1 (1)
Vertebral artery dissection (Nervous system disorders) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ectopic pregnancy with contraceptive device (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Embedded device (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levonorgestrel IUS (Mirena, BAY86-5028) (N=362)
Bacterial vaginosis (Infections and infestations) | 27 (40)
Nasopharyngitis (Infections and infestations) | 21 (29)
Urinary tract infection (Infections and infestations) | 27 (35)
Weight increased (Investigations) | 33 (33)
Anxiety (Psychiatric disorders) | 20 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT02985541/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT02985541/SAP_001.pdf